CLINICAL TRIAL: NCT05304156
Title: Single-cell Dynamic Profiling in Adults With Newly Diagnosed Acute Myeloid Leukemia Treated With Intensive Chemotherapy. A THEMA Study"
Acronym: DYNHAEMICS
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP 211175
Record Dates: First submitted 2022-01-28; First posted 2022-03-31 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Standard of Care in patients with AML: Standard of Care including a first course containing one of the following backbones without addition of third agent before day 8 of induction (approved drugs such as midostaurine or investigational agents administered beyond day 8 are allowed) :
  * 7+3 induction 3+7 with daunorubicin (or idarubicin) and cytarabine
  * CPX-351 induction
  Interventions: Other: Biobanking blood and bone marrow specimens

INTERVENTIONS:
Other: Biobanking blood and bone marrow specimens — Interventions, procedures added for research purposes :
  Blood Samples :
  * Peripheral blood (20mL EDTA) (at Screening, pre-ICT Day 1, Day1 H8, Day 2, Day 3, Day 4 and Day of EOI evaluation
  Bone Marrow samples :
  * Biopsy at Screening and at EOI Evaluation
  * Additional volume (2mL EDTA) on the Screening,2 and EOI Evaluation aspirations for single-cell analyses.
  * Aspiration at D8 for Smears and 2 mL EDTA for single-cell analyses (instead of D15 standard care).

SUMMARY:
The detailed molecular and cellular mechanisms underpinning the clinical activity of most chemotherapies in cancers remain incompletely understood. Understanding how these drugs really act is a prerequisite for their rational therapeutic optimization.

Recent observations suggest that early molecular and cellular changes in cancer cells upon chemotherapy exposure may dictate their long-term fate.

We aim to address this question in previously untreated adult Acute Myeloid Leukemia (AML) patients treated with anthracycline/cytarabine association (either as free drugs, '7+3' regimen, or in liposomal formulation, CPX-351) by sequentially sampling peripheral blood during the first course of therapy, and by performing an early bone marrow reassessment. We will apply single cell RNA sequencing and multiparameter flow cytometry to correlate dynamic phenotypic landscapes with clinical outcomes (remission achievement and relapse-free survival).

The study will be carried in two phases. First, a feasibility phase will be carried in the first 20 patients irrespective of the genetic make-up of their leukemic cells to identify the optimal pre-analytical conditions for single-cell transcriptional profiling.

Second, an expansion phase will be carried focusing on two genetically subsets of patients chosen on the basis of their relative abundance and variability of clinical outcome, namely NPM1c-mutated AML (30% of patients, 60% cure rate) and NPM1-wildtype intermediate-risk AML (25% of patients, 40% cure rate), to correlate single-cell fates with remission and with long-term remission-free survival.

ELIGIBILITY:
Inclusion Criteria:

* aged ≥18 years old,
* have a newly diagnosed AML according to WHO criteria

  o patients with AML related to prior chemotherapy or radiotherapy for another cancer will be eligible,
* have signed the informed consent form of the e-THEMA observatory trial
* have ≥10% blasts (blasts+myeloblasts) on the peripheral blood smear at screening,
* have ≥20% blasts on the bone marrow smear at screening,
* have not received any treatment for AML except for hydroxyurea and/or 6-mercaptopurine and steroids

  o Patients having previous treatments for antecedent myeloid neoplasms including hypomethylating agents remain eligible,
* Eligible to intensive chemotherapy, due to general health status,
* ECOG performance status ≤ 2,
* Patient is planned to receive anthracycline (daunorubicin [DNR] or idarubicine [IDA]) - cytarabine 7+3 with or without gemtuzumab ozogamycin (GO) or midostaurine, or CPX-351 as first induction course,
* Weighing 50 kg or more (compliance to Loi Jardé for PB sampling),
* Written informed consent obtained prior to any screening procedures,
* Eligible for National Health Insurance in France.

Exclusion Criteria:

* Suspected or proven acute promyelocytic leukemia based on morphology, karyotype or molecular assay,
* Failure to perform bone marrow aspiration at diagnosis,
* Unstable angina, New York Heart Association (NYHA) class 3 or 4 congestive heart failure,
* Prior anthracycline exposure more than 360 mg/m²,
* Previous therapy for AML with any other investigational agent or cytotoxic drug, within 28 days before starting treatment. Only hydroxyurea is permitted for the control of blood counts. Treatments for an antecedent myeloid neoplasm (MDS or MPN) are not considered as exclusion criteria.
* Women who are pregnant or breastfeeding.
* Any of concurrent severe and/or uncontrolled medical condition, which could compromise participation in the study.
* Enrolment in a clinical trial which could compromise participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients already included in eTHEMA observationnal cohort
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-04-26 (Actual); Primary Completion 2026-04-26 (Estimated); Study Completion 2026-05-26 (Estimated)

PRIMARY OUTCOMES:
Successful single-cell RNA-Seq (sc-RNA-Seq) assesment | up to 8 days
  Successful sc-RNA-Seq assessment is defined as the detection of > 1000 cells representing > 50% of the total number of viable loaded cells, with > 1000 reads per cell
Complete Remission (CR) without MRD | End of induction (day 28 to day 56)

SECONDARY OUTCOMES:
Event-Free Survival | at 5 years
Cumulative Incidence of Relapse | at 5 years
Overall Survival | at 5 years

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Hôpital Avicenne, Bobigny
  - Hôpital Saint Louis, Paris

IPD SHARING:
Plan to Share IPD: Undecided